CLINICAL TRIAL: NCT03787550
Title: Pharmacokinetics/Pharmacodynamics of the Sedatives, Analgesics and Antibiotics in Patients Receiving Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: PK/PD of the Sedatives, Analgesics and Antibiotics in Patients Receiving ECMO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECMO001
Record Dates: First submitted 2018-11-21; First posted 2018-12-26 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-05

CONDITIONS: Drug Effect
Keywords: ECMO; Sedatives; Analgesics; Antibiotics
MeSH Terms: interventions — Analgesics; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Model building group: The data from the patients in the model building group will be used to build the population PK/PD model. Two to six blood samples will be collected during at least one dose interval at the steady-state, including one sample from the start of ECMO and one at the end of ECMO.
  Interventions: Drug: The Sedatives, analgesics and antibiotics
- Model validation group: The data from the patients in the model building group will be used to build the population PK/PD model. Two to three blood samples will be collected during at least one dose interval at the steady-state, including one sample from the start of ECMO and one at the end of ECMO.
  Interventions: Drug: The Sedatives, analgesics and antibiotics

INTERVENTIONS:
Drug: The Sedatives, analgesics and antibiotics — The sedatives (dexmedetomidine, midazolam, propofol), analgesics (butorphanol, remifentanil, sufentanil), and six antibiotics (linezolid, voriconazole, tigecycline, teicoplanin, caspofungin and meropenem) will be used according to the clinical need.

SUMMARY:
It is a multi-center, open-label, observational study aimed to understand the pharmacokinetics and pharmacodynamics of the commonly used sedative, analgesic and antibiotic drugs in adult patients supported with extracorporeal membrane oxygenation (ECMO), by measuring the plasma concentrations and the clinical effect of dexmedetomidine, midazolam, butorphanol, remifentanil, sufentanil, propofol, linezolid, tigecycline, teicoplanin, caspofungin, voriconazole and meropenem.

ELIGIBILITY:
Inclusion Criteria:

* Patient given the sedatives, analgesics and antibiotics of interest during ECMO.
* Age from 18 to 85 years old.
* Multiple blood sampling is acceptable.

Exclusion Criteria:

* Patients who are allergic to the investigated drugs.
* Patients who are pregnant.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients undergoing ECMO will be invited to participate. At least 2-12 subjects will be enrolled to build a pharmacokineic model for each drug, and 1-4 subjects for external validation for each drug. The investigators plan to study the sedatives, analgesics and antibiotics with the initial sample size at 36 in total.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2020-02-07 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Minimum Plasma Concentration [Cmin] | Up to 24 hours.
  The minimum plasma concentration (the trough concentration), usually collected before the next dose.
Area Under the Curve [AUC] | Up to 24 hours.
  The area under the curve during the dose interval. It also can be calculated by the dose and the clearance of the drug.
Maximum Plasma Concentration [Cmax] | Up to 24 hours.
  The maximum plasma concentration, usually at the end of the infusion during an dose interval.

SECONDARY OUTCOMES:
ICU mortality | Up to 60 days.
  The intensive care unit (ICU) mortality is calculated as the number of deaths of the enrolled patients admitted to the ICU, divided by the number of the enrolled patient discharges from the ICU (including deaths and transfers), and often presented as percentage.
Hospital mortality | Up to 60 days.
  The hospital mortality is calculated as the number of deaths of the enrolled patients divided by the number of the total enrolled patient, and often presented as percentage.
Mechanical ventilation duration | Up to 60 days.
  Mechanical ventilation duration is the length of days the patients on the mechanical ventilation.
ICU length of stay (LOS) | Up to 60 days.
  ICU length of stay (LOS) is the length of days the patients in the ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Chunbo Chen, Ph. D., Study Chair — Guandong General Hospital
Locations (3):
- China (3):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong